CLINICAL TRIAL: NCT01130597
Title: A Multicenter, Open-Label, Single-Arm Study to Evaluate a Titration Regimen for Patiromer in Heart Failure Patients With Chronic Kidney Disease
Brief Title: Evaluation of Patiromer Titration in Heart Failure Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RLY5016-204
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2015-12

CONDITIONS: Heart Failure
Keywords: HF; Heart failure; hyperkalemia; chronic kidney disease; prevention of hyperkalemia in heart failure participants
MeSH Terms: conditions — Heart Failure; Hyperkalemia; Renal Insufficiency, Chronic | interventions — patiromer; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patiromer (Experimental): spironolactone + patiromer
  Interventions: Drug: patiromer; Drug: spironolactone

INTERVENTIONS:
Drug: patiromer — Active investigational drug
  Other Names: RLY5016; Veltassa
Drug: spironolactone

SUMMARY:
The purpose of this study was to evaluate the feasibility of individualized titration of patiromer according to serum potassium. This study also assessed the safety and tolerability of patiromer and the effects of patiromer on serum potassium in heart failure (HF) participants with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
This was an open-label, single-arm study to evaluate a titration regimen for patiromer in approximately 63 HF participants with CKD receiving one or more of the following: angiotensin-converting enzyme inhibitors (ACEIs), angiotensin II receptor blockers (ARBs), or beta blockers (BBs). This study was considered to be exploratory.

Upon successful completion of screening evaluations (-10 to -5 days prior to enrollment), all eligible participants were assigned at Baseline (Day 0 visit) to an initial dose of patiromer (20 g/day) and spironolactone (25 mg/day).

Study visits for enrolled participants were scheduled for Days 3, 7, 14, 21, 28, 35, 42, 49 and 56. A follow-up visit occurred on Day 63.

At selected study visits, patiromer or spironolactone doses may have been titrated. The study dosing algorithm was designed to maintain an individual's serum potassium value in the range of 4.0 - 5.1 mEq/L (based on local lab data).

Any participant with a local laboratory serum potassium value < 3.5 or > 5.5 mEq/L on two consecutive scheduled study visits, despite titration of patiromer or spironolactone, were withdrawn from the study, permanently discontinued patiromer and spironolactone, and returned for a follow-up visit within 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HF clinically indicated to receive spironolactone therapy
2. Age 18 years or older
3. Local laboratory serum potassium values of 4.3 - 5.1 mEq/L at screening and baseline
4. CKD (estimated glomerular filtration rate [eGFR] < 60 mL/min/1.73m2 at screening based on central lab creatinine measurement)
5. On at least one of the following HF therapies: ACEI, ARB, or BB
6. Females of child-bearing potential must be non-lactating, must have a negative serum pregnancy test at screening, and must have used a highly effective form of contraception for at least 3 months before study drug administration, during the study, and for one month after study completion
7. Male participants and/or their female partners of child-bearing potential must use a highly effective form of contraception during the study and for 3 months after study completion
8. Provide their written informed consent prior to participation in the study

Exclusion Criteria:

1. History of bowel obstruction, swallowing disorders, severe gastrointestinal disorders or major gastrointestinal surgery
2. Uncorrected primary severe valvular disease, known obstructive or restrictive cardiomyopathy, uncontrolled or hemodynamically unstable arrhythmia
3. Coronary-artery bypass graft, percutaneous intervention (e.g., cardiac, cerebrovascular, aortic), or major surgery including thoracic and cardiac, within 3 months prior to baseline or anticipated need during study participation
4. Heart transplant recipient, or anticipated need for transplant during study participation
5. Any of the following events having occurred within 2 months prior to baseline: unstable angina as judged by the Investigator, unresolved acute coronary syndrome, transient ischemic attack or stroke
6. Current dialysis participant, or anticipated need for dialysis during study participation
7. Prior kidney transplant, or anticipated need for transplant during study participation
8. Metastatic, late-stage or end-stage cancer with < 12 months life expectancy or at risk for tumor lysis syndrome
9. History of alcoholism or drug/chemical abuse within 1 year
10. Sustained systolic blood pressure > 180 or < 90 mmHg
11. Liver enzymes [alanine aminotransferase (ALT), aspartate aminotransferase (AST)] > 3 times upper limit of normal
12. Loop and thiazide diuretics that have not been stable for at least 21 days prior to baseline or not anticipated to remain stable during study participation
13. Use of any intravenous cardiac medications within 21 days prior to baseline, or their anticipated need during study participation
14. Current use of polymer-based drugs (e.g., sevelamer, sodium polystyrene sulfonate, colesevelam, colestipol), phosphate binders (e.g., lanthanum carbonate), or other potassium binders, or their anticipated need during study participation
15. Use of potassium sparing medication including aldosterone antagonists or potassium supplements in the last 21 days prior to baseline
16. Use of any investigational medication within 30 days or 5 half-lives, whichever is longer, prior to baseline
17. Participants who have taken investigational product in this study, or a previous patiromer study
18. Inability to consume the study medication, or, in the opinion of the Investigator, inability to comply with the protocol
19. In the opinion of the Investigator, any medical condition, uncontrolled systemic disease, serious intercurrent illness, or extenuating circumstance occurring or persisting, within 30 days prior to baseline, that would significantly decrease study compliance or jeopardize the safety of the participant or affect the validity of the trial results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Operations, Study Director — Relypsa, Inc.
Locations (13):
- Georgia (8):
  - Investigator Site 11, Tbilisi
  - Investigator Site 12, Tbilisi
  - Investigator Site 13, Tbilisi
  - Investigator Site 14, Tbilisi
  - Investigator Site 15, Tbilisi
  - Investigator Site 16, Tbilisi
  - Investigator Site 17, Tbilisi
  - Investigator Site 18, Tbilisi
- Slovenia (5):
  - Investigator Site 25, Golnik
  - Investigator Site 27, Izola
  - Investigator Site 21, Ljubljana
  - Investigator Site 22, Maribor
  - Investigator Site 26, Slovenj Gradec

REFERENCES:
- [Derived] Pitt B, Bushinsky DA, Kitzman DW, Ruschitzka F, Metra M, Filippatos G, Rossignol P, Du Mond C, Garza D, Berman L, Lainscak M; Patiromer-204 Investigators. Evaluation of an individualized dose titration regimen of patiromer to prevent hyperkalaemia in patients with heart failure and chronic kidney disease. ESC Heart Fail. 2018 Jun;5(3):257-266. doi: 10.1002/ehf2.12265. Epub 2018 Jan 25. PMID 29369537

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were ≥ 18 years old, had a history of chronic HF, were clinically indicated to initiate spironolactone therapy, had a serum potassium measurement of 4.3 - 5.1 mEq/L at screening and baseline, had CKD (eGFR < 60 mL/min/1.73 m2 at screening), and were taking one or more HF therapies (ACEIs, ARBs, or BBs).
Groups:
- Patiromer: Spironolactone + Patiromer
  Participants received patiromer (20 g/day, administered as a divided dose of 10 g in the morning and 10 g in the evening) and spironolactone (25 mg/day, administered once daily), orally. After Day 3, at the first occurrence of a serum potassium value of ≤ 5.1 mEq/L, the spironolactone dose was increased once to 50 mg/day; dose reductions were not allowed.
Period: Overall Study
Arm/Group | Patiromer
Started | 63
Completed | 56
Not Completed | 7
Not completed — Protocol-specified (High K+) | 1
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patiromer
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 46
Age, Continuous [Mean (Full Range); unit: years] | 70.8 [53 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Potassium in the Range of 3.5 - 5.5 mEq/L at the End of Treatment
Time Frame: 56 days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 63
percentage of participants | 90.5
Statistical Analysis 1: Comparison: Patiromer; Test type: Superiority or Other; Percentage of Participants = 90.5, 95% CI 2-sided [80.4 to 96.4] — Clopper-Pearson was used to arrive at the 95% Confidence Interval

2. Secondary Outcome: Percentage of Participants With Serum Potassium in the Range of 3.5 - 5.5 mEq/L at Week 4
Time Frame: 28 Days
Population: Participants with available data at Week 4.
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 61
percentage of participants | 96.7

3. Secondary Outcome: Percentage of Participants With Serum Potassium in the Range of 3.5 - 5.5 mEq/L at Week 8
Time Frame: 56 Days
Population: Participants with available data at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 57
percentage of participants | 93.0

4. Secondary Outcome: Percentage of Participants With Serum Potassium in the Range of 4.0 - 5.1 mEq/L at Week 4
Time Frame: 28 Days
Population: Participants with available data at Week 4.
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 61
percentage of participants | 78.7

5. Secondary Outcome: Percentage of Participants With Serum Potassium in the Range of 4.0 - 5.1 mEq/L at Week 8
Time Frame: 56 Days
Population: Participants with available data at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 57
percentage of participants | 86.0

6. Secondary Outcome: Percentage of Participants With Serum Potassium in the Range of 4.0 - 5.1 mEq/L at the End of Treatment
Time Frame: 56 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 63
percentage of participants | 84.1
Statistical Analysis 1: Comparison: Patiromer; Test type: Superiority or Other; Percentage of Participants = 84.1, 95% CI 2-sided [72.7 to 92.1] — Clopper-Pearson was used to arrive at the 95% Confidence Interval

7. Secondary Outcome: Mean Dose of Patiromer at End of Treatment
Time Frame: 56 Days
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Patiromer
Number analyzed (Participants) | 63
grams | 22.5 (7.8)

8. Secondary Outcome: Percentage of Participants Requiring Patiromer Uptitration
Time Frame: 56 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 63
percentage of participants | 33.3

9. Secondary Outcome: Percentage of Participants Requiring Patiromer Downtitration
Time Frame: 56 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 63
percentage of participants | 12.7

10. Secondary Outcome: Median Time to First Patiromer Dose Titration
Time Frame: 56 Days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Patiromer
Number analyzed (Participants) | 63
days | 21 [14.0 to 36.0]

11. Secondary Outcome: Mean Number of Patiromer Titrations
Time Frame: 56 Days
Measure: Mean (Standard Deviation); unit: patiromer titrations
Arm/Group | Patiromer
Number analyzed (Participants) | 63
patiromer titrations | 1.3 (1.1)

12. Secondary Outcome: Mean Patiromer Dose at Week 1
Time Frame: Up to Week 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Patiromer
Number analyzed (Participants) | 63
grams | 20.0 (0.0)

13. Secondary Outcome: Mean Patiromer Dose at Week 4
Time Frame: Up to Week 4
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Patiromer
Number analyzed (Participants) | 63
grams | 21.9 (8.5)

14. Secondary Outcome: Mean Patiromer Dose at Week 8
Time Frame: Up to Week 8
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Patiromer
Number analyzed (Participants) | 63
grams | 23.0 (12.4)

15. Secondary Outcome: Mean Change From Baseline in Serum Potassium to End of Treatment
Time Frame: 56 Days
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Patiromer
Number analyzed (Participants) | 63
mEq/L | -0.13 (0.686)

16. Secondary Outcome: Percentage of Participants Discontinuing Due to Hyperkalemia (Serum Potassium > 5.5 mEq/L)
Time Frame: 56 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 63
percentage of participants | 1.6

17. Secondary Outcome: Percentage of Patients Whose Spironolactone Dose Was Increased Up to 50 mg/Day
Time Frame: 56 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer
Number analyzed (Participants) | 63
percentage of participants | 100

18. Secondary Outcome: Change in Urine Albumin to Creatinine Ratio (ACR) From Baseline to Week 4 Among Participants With ACR ≥ 30 mg/g at Baseline
Time Frame: Baseline and Day 28
Population: Participants with urine ACR ≥ 30 mg/g at baseline and available data at Week 4
Measure: Mean (Standard Error); unit: mg/g
Arm/Group | Patiromer
Number analyzed (Participants) | 31
mg/g | -291.01 (130.7973)

19. Secondary Outcome: Change in ACR From Baseline to Week 8 Among Participants With Urine ACR ≥ 30 mg/g at Baseline
Time Frame: Baseline and Day 56
Population: Participants with urine ACR ≥ 30 mg/g at baseline and available data at Week 8
Measure: Mean (Standard Error); unit: mg/g
Arm/Group | Patiromer
Number analyzed (Participants) | 30
mg/g | -291.06 (141.5644)

ADVERSE EVENTS:
Time Frame: Up to 7 days after Day 56 or last patiromer dose, whichever was earlier.
Description: Participants who received at least one dose of trial medication.
Arm/Group | Patiromer
Serious Adverse Events (participants affected / at risk) | 6/63
Other Adverse Events (participants affected / at risk) | 4/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer (N=63)
Acute myocardial infarction (Cardiac disorders) | 1
Sudden cardiac death (General disorders) | 1
Sudden death (General disorders) | 1 — Sudden death occurred during the follow up period, after completing the study.
Pneumonia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer (N=63)
Abdominal discomfort (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements generally provide that PI cannot publish single site data before publication of the multi-site publication, unless 1 year has elapsed since completion of the study at all sites. Thereafter, PI may publish provided that PI shall: provide a copy of the publication to sponsor at least 60 days in advance of submission for publication; delete sponsor's confidential information as requested; and delay publication up to an additional 90 days to permit protection of intellectual property.